CLINICAL TRIAL: NCT00414999
Title: A Phase 1, Double-Masked, Placebo-Controlled, Dose-Escalation Study (in Two Parts) of TG100801 and a Colored Vehicle in Adult Healthy Volunteers
Brief Title: A Phase 1 Safety Study of TG100801 Eye Drops in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TargeGen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPH-TG100801-001
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2007-07

CONDITIONS: Macular Degeneration; Diabetic Retinopathy
Keywords: Macular degeneration; Vascular diseases; Retinal disorders; Macular edema
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Vascular Diseases; Retinal Diseases; Macular Edema | interventions — 4-chloro-3-(5-methyl-3-((4-(2-pyrrolidin-1-ylethoxy)phenyl)amino)-1,2,4-benzotriazin-7-yl)phenol

INTERVENTIONS:
Drug: TG100801

SUMMARY:
The formation of new blood vessels (angiogenesis), blood vessel leakage, and inflammation contribute to the progression of the eye disease, age-related macular degeneration (AMD), which is the leading cause of irreversible, severe loss of vision in people 55 years of age and older in the developed world. TG100801 is a new drug that inhibits ocular angiogenesis, vascular leak, and inflammation in laboratory studies, and may have great utility in the treatment of diseases such as AMD.

The purpose of this study is to assess the safety, ocular tolerability, and blood pharmacokinetics of TG100801 at escalating doses in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Male or female healthy volunteers who meet the following criteria are eligible for inclusion in the study. Subjects who participate in Part A of the study may not participate in Part B.

* Age > 18 years (50% of subjects must be > 40 years of age).
* Corrected visual acuity > 20/25 in both eyes.
* Intraocular pressure (IOP) < 21 mm Hg, with a difference between eyes of < 4 mm Hg.
* Ability to tolerate and self-administer vehicle eye drops to the satisfaction of study staff.
* Tolerance of a commercially available benzalkonium chloride-preserved, artificial tear solution in one eye.
* Normal slit lamp exam and dilated fundoscopic exam within 2 weeks of dosing.
* Normal clinical laboratory profiles, defined as complete blood count, serum chemistry, and urinalysis values within the normal range.
* Willing to abstain from the concomitant use of ocular or systemic medication (excluding acetaminophen and multivitamins) from 2 weeks prior to start of study dosing until study completion.
* Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other study-related procedures.
* Provide written informed consent to participate.

Exclusion Criteria:

Subjects who meet any of the following criteria are excluded from the study:

* History of ocular surgery, trauma, or chronic ocular disease.
* Current use of contact lenses or discontinuation of contact lens use within 2 weeks of the first dosing day.
* Any ocular abnormalities or ocular symptoms (defined as a non-zero score on assessment scales).
* Use of ocular agents (including eye drops) within the past 2 months or anticipated use of ocular agents during the study period.
* Systemic corticosteroid use within the past 6 months.
* History or evidence of ocular infection, inflammation, blepharitis, or conjunctivitis with 2 months; history of herpes simplex keratitis.
* Presence of a nonhealing wound, ulcer, fracture, or any medical condition associated with bleeding.
* Use of antimitotic or antimetabolite therapy within 2 months of enrollment.
* Loss, donation, or removal of 400 mL or more of blood within the past 2 months.
* Women who are pregnant or breastfeeding, or nonsterile or premenopausal women who refuse to use two proven methods of contraception during and for at least 2 weeks following the final dose of study drug.
* Enrollment in another investigational drug or device study within 2 months of study entry.
* Ongoing cardiac arrhythmias or prolongation of the QTc interval to > 450 msec for males or > 470 msec for females.
* Known liver, kidney, cardiovascular, neurologic, or pulmonary disease; treated or untreated hypertension; current or history of drug or alcohol abuse.
* Known human immunodeficiency virus- or acquired immunodeficiency syndrome-related illness.
* Known intolerance to any excipients in the study drug formulation.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, would affect the subject's ability to follow study-related procedures, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Part A: Safety & tolerability of vehicle & 2 concentrations of TG100801 (ophthalmic examinations, ocular comfort ratings, ocular/systemic adverse events, lab tests) when administered twice a day for 1 day, assessed up to 5 (+/- 1) days following dosing.
Part B: Safety & tolerability of 2 concentrations of TG100801 (ophthalmic examinations, ocular comfort ratings, ocular/systemic adverse events, lab tests) when administered twice a day for 14 days, assessed up to 7-14 days following dosing.

SECONDARY OUTCOMES:
Systemic pharmacokinetics (Part B only)

CONTACTS AND LOCATIONS:
Overall Officials: Philip T Leese, M.D., Principal Investigator — Quintiles Phase One Services, Inc.
Locations (1):
- Quintiles Phase One Services, Inc., Lenexa, Kansas, United States

REFERENCES:
- See also: American Macular Degeneration Foundation — http://www.macular.org